CLINICAL TRIAL: NCT01308489
Title: Comparison of Minimally Invasive Approaches of Spine Tumor Surgery
Brief Title: Minimally Invasive Surgery in Treating Patients With Spinal Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject response
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10115; NCI-2011-00231 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-03-01; First posted 2011-03-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Adult Spinal Cord Neoplasm; Recurrent Adult Spinal Cord Neoplasm; Spinal Bone Metastases; Spinal Cord Metastases
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (posterior spinal tumor resection) (Experimental): Patients undergo posterior spinal tumor resection on day 0.
  Interventions: Procedure: therapeutic conventional surgery; Procedure: quality-of-life assessment
- Arm II (anterior and posterior spinal tumor resection) (Experimental): Patients undergo anterior and posterior tumor resection on day 0.
  Interventions: Procedure: therapeutic conventional surgery; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo posterior spinal tumor resection
  Arms: Arm I (posterior spinal tumor resection)
Procedure: therapeutic conventional surgery — Undergo anterior and posterior spinal tumor resection
  Arms: Arm II (anterior and posterior spinal tumor resection)
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This randomized clinical trial studies minimally invasive surgery in treating patients with spinal tumors. Posterior spinal tumor resection and anterior and posterior spinal tumor resection are less invasive types of surgery for spinal tumors and may have fewer side effects and improve recovery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Length of operation (operating room [OR] time). II. Estimated blood loss (EBL). III. Complication rate. IV. Neurological preservation.

SECONDARY OBJECTIVES:

I. Motor strength and sensory level (neurological outcome). II. Bladder and bowel function. III. Post-operative pain. IV. Hospital length of stay (recovery time). V. Arthrodesis.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo posterior spinal tumor resection on day 0.

ARM II: Patients undergo anterior and posterior spinal tumor resection on day 0.

After completion of study treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of primary, secondary or metastatic spine tumor and be undergoing any posterior spinal fusion with or without anterior fusion anywhere from occiput to sacrum
* Greater than 3 month life expectancy
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients who are not surgical candidates for spine tumor removal, determined by the surgical team
* Patients who have undergone previous spine surgery for tumor removal will be excluded
* Patients with renal cell carcinoma
* As there is an emphasis on blood loss and length of surgery, the critical variable for homogeneity is the vascularity of the tumor; hypervascular spine tumors are regarded by surgeons as amongst the most challenging of cases; by far the three most common hypervascular metastatic tumors are those arising from renal cell carcinoma, thyroid carcinoma and melanoma; these pathologies are usually regarded as a distinct subset for this reason in the majority of studies; because we rarely encounter the later two pathologies in our practice, we chose to include only the former; however, to further homogenize our study population we will exclude all three of the known hypervascular metastatic spine tumors
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Estimated blood loss (EBL); in milliliters (ml) | Day 0
  Will be comparing means with the Wilcoxon test.
Length of operation (OR time) | Day 0
  Will be comparing means with the Wilcoxon test.
Complication rate | Day 0
Neurological preservation | Post operation day 90

SECONDARY OUTCOMES:
Length of stay | Less than 7 days
Pain symptoms | Pre-operation, post-op day 3, discharge, post-op days 7, 28, 60, and 90
Assessment of neurologic function using the ASIA (American Spinal Injury Association) Impairment Scale | Pre-operation, post-op day 3, discharge, post-op days 7, 28, 60, and 90
  This is an assessment of sensory and motor functions based upon the ASIA Impairment Scale
Evaluation of arthrodesis | Post-op day 1, 28, and 90
  Plain x-ray films and CT scans are used to determine the success of arthrodesis (spinal fusion in this case) which is the artificial induction of joint ossification between two bones via surgery. This is done to relieve intractable pain in a joint which cannot be managed by pain medication.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Jandial, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States